CLINICAL TRIAL: NCT05633095
Title: A Prospective Pilot Study to Evaluate Efficacy and Safety of Medical Device-Neuclare in Patient With Mild Cognitive Disorder and Early Dementia
Brief Title: The Pilot Study of Medical Device-Neuclare for Patients With Mild Cognitive Disorder and Early Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deepsonbio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Deepsonbio_Neuclare
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-11

CONDITIONS: Dementia, Mild; Cognitive Disorder Mild
MeSH Terms: conditions — Dementia; Lymphoma, Follicular; Neurocognitive Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The patient with mild cognitive disorder and early dementia who will be treated with the medical device-Neuclare
  Interventions: Device: Neuclare

INTERVENTIONS:
Device: Neuclare — It is used to stimulate the brain for a certain period of time to improve cognitive impairment in patients with cognitive disorder. In this clinical trial, it is used for patients with mild cognitive disorder and demincia symptoms.

SUMMARY:
This clinical trial aims to explore the effectiveness and safety of cognitive function improvement of Neuclare, a science medical device, for patients with mild cognitive impairment and early Alzheimer's disease.

Through methods such as Trail Making Test Black & White, Attention Questionnaire Scale(AQS), Neuropsychiatric Inventory (NPI), etc, cognitive function improvement before and after using Neuclare will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 to 90
* Patients who meet "Probable Alzheimer's disease" and "Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV)" criteria for dementia
* Patients with CDR (clinical dementia rating) from 0.5 to 1 and MMSE-II over 18
* Upon hearing and fully understanding the detailed explanation of this clinical trial, a person who has voluntarily decided to participate and agreed in writing to comply with the precautions

Exclusion Criteria:

* Patient with pathological lesions in the brain identified by MRI
* Patients with metabolic disorders such as thyroid dysfunction, hyperglycemia, hypoglycemia, liver or kidney dysfunction, and long-term use of drugs that will cause cognitive decline (e.g., anticholinergic drugs)
* History of epileptic seizures or depression or psychiatric abnormalities or with visual acuity and fluctuations in cognitive decline
* History of psychiatric disorder other than the inclusion criteria.
* A person with a severe history of cancer/tuberculosis
* A person who has or is taking psychiatric or peripheral/central nervous system drugs
* A person who has contact dermatitis or sensitive skin abnormalities
* Patients with a high fever of 40 degrees or higher based on eardrum body temperature
* A person whose bleeding is identified within the last 3 months due to a common procedure/surgery that may affect vital signs
* A person who is unable to perform MRI tests
* Pregnant women
* Patient with calcification in the brain identified by CT
* Patient with allergic to contrast agents such as Definity or Gadovist
* Other cases where the investigator judged that it is difficult to participate in the study;

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Change of Trail Making Test Black & White Score : From Baseline to Week 5 | Week 5
  Compare with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as evaluated by Trail Making Test Black & White Score

SECONDARY OUTCOMES:
Change of Attention Questionnaire Scale : From Baseline to Week 5 | Week 5
  Compare with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as evaluated by Attention Questionnaire Scale
Change of Neuropsychiatric Inventory Score : From Baseline to Week 5 | Week 5
  Compare with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as evaluated by Neuropsychiatric Inventory score
Change of Quality of life-AD Score : From Baseline to Week 5 | Week 5
  Compare with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as evaluated by Quality of life-AD Score
Change of MMSE-II Score : From Baseline to Week 5 | Week 5
  Compare with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as evaluated by MMSE-II Score
change of beta-amyloid deposition measured by Amyloid PET-CT : From Baseline to Week 5 | Week 5
  change of beta-amyloid deposition with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as measured by Amyloid PET-CT
Change of glucose metabolic rate in brain measured by FDG PET-CT : From Baseline to Week 5 | Week 5
  Compare glucose metabolic rate with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as measured by FDG PET-CT
Change of Aβ oligomer density measured by MDS-OAβ test result : From Baseline to Week 5 | Week 5
  Compare Aβ oligomer density with before and after using Neuclare for the treatment of mild cognitive disorder and early dementia as measured by MDS-OAβ test

CONTACTS AND LOCATIONS:
Overall Officials: SangYun Kim, M.D. ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No